CLINICAL TRIAL: NCT06542705
Title: Effect of Internal Brace on Outcomes Following ACL Reconstruction With Bone Patellar Bone (BTB) Autograft: A Randomized Controlled Trial
Brief Title: Effect of Internal Brace on Outcomes Following ACL Reconstruction With BTB Autograft
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 24-00423
Record Dates: First submitted 2024-08-05; First posted 2024-08-07 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: ACL Reconstruction

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Internal Brace (Experimental): Patients will undergo ACL Reconstruction (ACLR) with an internal brace. Patients will undergo standard perioperative protocol and be followed at typical time points after surgery (2 weeks, 6 weeks, 3 months, 6 months, 12 months). At 12 months postoperative, a follow-up MRI will be obtained to evaluate healing and at 12 months and 24 months follow up KT-1000 testing will be conducted.
  Interventions: Device: Arthrex Internal Brace; Procedure: ACL Reconstruction
- Standard ACLR (Active Comparator): Patients will undergo ACLR without an internal brace. Patients will undergo standard perioperative protocol and be followed at typical time points after surgery (2 weeks, 6 weeks, 3 months, 6 months, 12 months). At 12 months postoperative, a follow-up MRI will be obtained to evaluate healing and at 12 months and 24 months follow up KT-1000 testing will be conducted.
  Interventions: Procedure: ACL Reconstruction

INTERVENTIONS:
Device: Arthrex Internal Brace — The Arthrex Internal Brace method for ACL reconstruction consists of suture tape used to reinforce the ACL during surgery. This suture tape is secured in place with bioabsorbable anchors that gradually degrade within the body over time.
  Other Names: AR-1593-BC
  Arms: Internal Brace
Procedure: ACL Reconstruction — All patients will undergo ACL reconstruction (ACLR) with or without an internal brace. ACLR technique will be standardized to standard anteromedial (AM) portal femoral drilling to ensure consistency between surgeons.

SUMMARY:
The purpose of this study is to assess Anterior Cruciate Ligament (ACL) healing through analyzing clinical, radiographic, functional and patient-reported outcomes following ACL reconstruction with bone-tendon-bone autograft with and without internal bracing.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing ACLR with BTB autograft
* Patients ages 18-35, inclusive
* Ability to undergo standard rehab protocol and full, painless range of motion at the time of surgery of their operative knee

Exclusion Criteria:

* Osteoarthritis defined by Kellgren-Lawrence grade 2 or higher on preoperative weightbearing radiographs
* Significant chondral injury as defined by grade 3-4 lesion greater than 2cm2
* History of autoimmune or inflammatory disease
* Prior ipsilateral knee ligament surgery or multi-ligament knee injury
* Concomitant Lateral extra-articular tenodesis (LET) procedure
* History of contralateral ACL surgery
* Younger than 18 years of age
* Older than 35 years of age

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-03-17 (Actual); Primary Completion 2029-03 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
Side to side difference in laxity as measured by the KT-1000 Arthrometer | Month 12 Post-Operation
  The KT-1000 knee arthrometer (KT-1000) is an objective instrument to measure anterior tibial motion relative to the femur for anterior cruciate ligament (ACL) reconstruction. The side-to-side differences comparing the injured and normal extremity allow the determination of a diagnosis of increased anterior-posterior laxity. A side-to-side difference of less than 3mm at 30lb and the manual maximum is considered normal. A side-to-side difference between 3 and 5mm is considered a grey area. A side-to-side difference of more than 5mm is considered diagnostic of an ACL tear.
Side to side difference in laxity as measured by the KT-1000 Arthrometer | Month 24 Post-Operation
  The KT-1000 knee arthrometer (KT-1000) is an objective instrument to measure anterior tibial motion relative to the femur for anterior cruciate ligament (ACL) reconstruction. The side-to-side differences comparing the injured and normal extremity allow the determination of a diagnosis of increased anterior-posterior laxity. A side-to-side difference of less than 3mm at 30lb and the manual maximum is considered normal. A side-to-side difference between 3 and 5mm is considered a grey area. A side-to-side difference of more than 5mm is considered diagnostic of an ACL tear.

SECONDARY OUTCOMES:
Pivot Shift Grade | Month 12 Post-Operation
  The Pivot Shift test is a dynamic, passive test to assess the rotational instability of the Anterior Cruciate Ligament in the knee.
  Pivot shift grades include: equal/0 (negative); glide/1; clunk/2; gross/3. A positive grade indicates injury to the Anterior Cruciate Ligament.
Pivot Shift Grade | Month 24 Post-Operation
  The Pivot Shift test is a dynamic, passive test to assess the rotational instability of the Anterior Cruciate Ligament in the knee.
  Pivot shift grades include: equal/0 (negative); glide/1; clunk/2; gross/3. A positive grade indicates injury to the Anterior Cruciate Ligament.
Change from Baseline in Visual Analogue Scale (VAS) - Pain Score at Month 12 Post-Operation | Baseline, Month 12 Post-Operation
  Participants rate their pain on a scale from 0 (no pain) to 10 (worst pain imaginable); the response is the total score.
Change from Baseline in Visual Analogue Scale (VAS) - Pain Score at Month 24 Post-Operation | Baseline, Month 24 Post-Operation
  Participants rate their pain on a scale from 0 (no pain) to 10 (worst pain imaginable); the response is the total score.
Change from Baseline in International Knee Documentation Committee (IKDC) Survey at Month 12 Post-Operation | Baseline, Month 12 Post-Operation
  This is a survey taken by patients to report how their knee is working for them. The IKDC is graded by adding the results and converting the result to a number on a scale from 0 to 100. Scores range from 0 (lowest level of function and highest level of symptoms) to 100 points (highest level of function and lowest level of symptoms).
Change from Baseline in International Knee Documentation Committee (IKDC) Survey at Month 24 Post-Operation | Baseline, Month 24 Post-Operation
  This is a survey taken by patients to report how their knee is working for them. The IKDC is graded by adding the results and converting the result to a number on a scale from 0 to 100. Scores range from 0 (lowest level of function and highest level of symptoms) to 100 points (highest level of function and lowest level of symptoms).
Change from Baseline in Lysholm Knee Scoring System Score at Month 12 Post-Operation | Baseline, Month 12 Post-Operation
  The Lysholm Knee Scoring System is an 8-item assessment of the prevalence of knee problems. The total score ranges from 0-100; scores between 95 and 100 are regarded as exceptional, 84 and 94 as acceptable, 65 to 83 as fair, and less than 65 as poor.
Change from Baseline in Lysholm Knee Scoring System Score at Month 24 Post-Operation | Baseline, Month 24 Post-Operation
  The Lysholm Knee Scoring System is an 8-item assessment of the prevalence of knee problems. The total score ranges from 0-100; scores between 95 and 100 are regarded as exceptional, 84 and 94 as acceptable, 65 to 83 as fair, and less than 65 as poor.
Tegner Activity Level Scale | Month 24 Post-Operation
  The Tegner activity level scale is a scale that aims to provide a standardized method of grading work and sporting activities. The Tegner activity level scale is a graduated list of activities of daily living, recreation, and competitive sports. The patient is asked to select the level of participation that best describes their current level of activity and that before injury.
  A score of 0 represents sick leave or disability pension because of knee problems, whereas a score of 10 corresponds to participation in national and international elite competitive sports. A score >6 can only be achieved if the person participates in recreational or competitive sport.

CONTACTS AND LOCATIONS:
Overall Officials: Michael J. Alaia, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset used in the published manuscript will be shared upon reasonable request beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research provided the investigator who proposes to use the data executes a data use agreement with NYU Langone Health. Requests may be directed to Michael.Alaia@nyulangone.org. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will be provided access upon reasonable request. Requests should be directed to Michael.Alaia@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.